CLINICAL TRIAL: NCT01750957
Title: A Randomized, Parallel Group, Double-Blind, Placebo-Controlled, Safety and Exploratory Efficacy and Pharmacokinetic, Study of RO4917523 in Pediatric Patients With Fragile X Syndrome
Brief Title: A Study of RO4917523 in Pediatric Patients With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP28571; 2011-004349-42 (EudraCT Number)
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO4917523 Dose A (Experimental)
  Interventions: Drug: RO4917523
- RO4917523 Dose B (Experimental)
  Interventions: Drug: RO4917523

INTERVENTIONS:
Drug: Placebo — orally daily, 12 weeks
  Arms: Placebo
Drug: RO4917523 — Dose A orally daily, 12 weeks
  Arms: RO4917523 Dose A
Drug: RO4917523 — Dose B orally daily, 12 weeks
  Arms: RO4917523 Dose B

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel-arm study will evaluate the safety and exploratory efficacy and pharmacokinetics of RO4917523 in pediatric patients with fragile X syndrome. Patients will be randomized to receive one of 2 dose levels of RO4917523 or placebo orally daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents, 5 to 13 years of age
* Diagnosis of fragile X syndrome based on prior DNA testing confirming Fragile X Mental Retardation 1 (FMR1) full mutation and qualifying scores on the ABC and CGI-S

Exclusion Criteria:

* Previous treatment with another mGlu5 receptor antagonist within the prior 3 months
* Participation in a clinical trial involving an investigational drug (unapproved) or non-drug treatment within the prior 6 weeks or 5 times the half-life (whichever is longer) before the start of this study
* Any uncontrolled, unstable clinically significant psychiatric condition other than fragile X syndrome
* History of suicidal behavior
* Other protocol defined inclusion/exclusion criteria may apply

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 15 weeks

SECONDARY OUTCOMES:
Efficacy: Neuropsychological/behavioral assessment scales (ADAMS/Clinical Global Impressions CGI-S, CGI-I/ GBAS/Aberrant Behavior Checklist ABC/Repeatable Battery for the Assessment of Neuropsychological Status RBANS/VAS behavior) | 15 weeks
Pharmacokinetics: Clearance (CL/F) | up to Week 12
Pharmacokinetics: Volume of distribution at steady-state (Vss/F) | up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- United States (20):
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Decatur, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Worcester, Massachusetts
  - Omaha, Nebraska
  - New York, New York
  - Cincinnati, Ohio
  - Media, Pennsylvania
  - Greenwood, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Seattle, Washington